CLINICAL TRIAL: NCT05609227
Title: Effect of a Mobile Application Developed for Hematopoietic Stem Cell Transplant Patients on Supportive Care Needs and Quality of Life
Brief Title: Effect of Mobile Application on Supportive Care Needs and Quality of Life Patients Undergoing Hematopoietic Stem Cell Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Baskent University (Other)
Collaborators: Ankara Oncology Research and Training Hospital (Network)
Responsible Party: Principal Investigator, Dila Başcı, MSc, Baskent University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: KA21/130
Record Dates: First submitted 2022-10-27; First posted 2022-11-08 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Hematologic Malignancy; Patient Education
Keywords: stem cell transplantation; mobile application; bone marrow transplant; quality of life; supportive care
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants will be stratified according to type of planned transplantation by preparatory outpatient clinic nurse; then will randomly assigned to two groups either intervention or control. The intervention group will get a mobile application developed compatible with IOS or android systems, containing information about the stem cell transplantation process, stem cell transplantation and nutrition, lifestyle recommendations, and answering possible questions of the patients and their relatives. The control group will receive standard care. The data of both groups will be collected on the first day of hospitalization, at controls during the first and third month.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mobile application (Experimental): Participants will get a mobile application containing information about information about all stages of stem cell transplantation process (pre, during and post).
  Interventions: Other: mobile application
- Control (No Intervention): Participants will receive routine care.

INTERVENTIONS:
Other: mobile application — The application, compatible with IOS and android systems for patients candidate for stem cell transplantation, could be applied whenever needed information relating to transplantation process.
  Arms: mobile application

SUMMARY:
The aim of this interventional study is to determine the effect of the mobile application on quality of life and supportive care in patient undergoing stem cell transplantation.The main questions it aims to answer are:

1. What is the effect of the education given with the mobile application on the quality of life of stem cell transplant patients?
2. What is the effect of the education given with the mobile application on supportive care of stem cell transplant patients?
3. What is the effect of the education given with the mobile application on anxiety levels of stem cell transplant patients? In the study, patients will be randomized into the group in which standard processes are applied and the group trained by the mobile application.

DETAILED DESCRIPTION:
Stem cell transplantation has been used for more than 50 years in the treatment of malignant and benign hematological diseases and some solid tumors. The stem cell transplant preparation process is a complex treatment that requires close follow-up in the hospital and after the transplant. Studies indicate that patients experience more intense worry and anxiety during the transplant process. Nursing care during the transplant period includes factors such as oral care, nutrition, mobilization, taking preventive measures against complications associated with neutropenia and thrombocytopenia, and these interventions have a positive effect on the patient's quality of life. Aim of this study is to determine the effect of the mobile application on quality of life and supportive care in patient undergoing stem cell transplantation. In the study, patients will be randomized into the group in which standard processes are applied and the group trained by the mobile application. Functional assessment scale (FACT-BMT), James Supportive Care and Needs Assessment Scale in Cancer Patients and Hospital Anxiety and Depression Scale were planned to be administered to both groups on the day of hospitalization and discharge day, and 3rd month follow up. The mobile application content will consist of 3 modules: information about the stem cell transplantation process, stem cell transplantation and nutrition, lifestyle recommendations, and answering possible questions of the patients and their relatives. At the end of the study, the test results of the patient groups will be compared both within themselves and with each other. The effects of standard and mobile application training on the test results of the patients and whether the results of the group receiving mobile application training differ from the standard training group will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing hematopoietic stem cell transplantation (autologous or allogeneic) for the first time
* Patients aged18 years or older,
* Patients able to communicate in Turkish as well as reading and writing.
* Those whose physical and mental conditions are suitable for participating in the research,
* Patients volunteered to participate in the study.

Exclusion Criteria:

* Being illiterate
* Patients not having a smartphone
* Patients not being able to use mobile application

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
quality of functionality | Baseline and 90th days
  Functional Assessment of Cancer Therapy-Bone Marrow Transplant (4th version) (Change from baseline to the 30th and 90th days will be assessed).
supportive care | Baseline and 90th days
  James Supportive Care Screening (Change from baseline to the 30th and 90th days will be assessed).
anxiety | Baseline and 90th days
  Distress thermometer (Change from baseline to the 30th and 90th days will be assessed).

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Abdurrahman Yurtaslan Ankara Onkoloji Eğitim ve Araştırma Hastanesi, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] Rozwadowski M, Dittakavi M, Mazzoli A, Hassett AL, Braun T, Barton DL, Carlozzi N, Sen S, Tewari M, Hanauer DA, Choi SW. Promoting Health and Well-Being Through Mobile Health Technology (Roadmap 2.0) in Family Caregivers and Patients Undergoing Hematopoietic Stem Cell Transplantation: Protocol for the Development of a Mobile Randomized Controlled Trial. JMIR Res Protoc. 2020 Sep 18;9(9):e19288. doi: 10.2196/19288. PMID 32945777
- [Background] Larson JL, Rosen AB, Wilson FA. The Effect of Telehealth Interventions on Quality of Life of Cancer Patients: A Systematic Review and Meta-Analysis. Telemed J E Health. 2018 Jun;24(6):397-405. doi: 10.1089/tmj.2017.0112. Epub 2017 Nov 7. PMID 29112484
- [Background] Moradian S, Voelker N, Brown C, Liu G, Howell D. Effectiveness of Internet-based interventions in managing chemotherapy-related symptoms in patients with cancer: a systematic literature review. Support Care Cancer. 2018 Feb;26(2):361-374. doi: 10.1007/s00520-017-3900-8. Epub 2017 Sep 25. PMID 28948360